CLINICAL TRIAL: NCT01030510
Title: The Effect of Remifentanil on the Onset Time of Rocuronium in Total Intravenous Anesthesia
Brief Title: Study of Rocuronium Onset Time According to Remifentanil Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: TIVA_rocu
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group R (Active Comparator): In group R, remifentanil was infused first before administrating propofol and rocuronium
  Interventions: Drug: the order of drug administration
- group P (Active Comparator): in group P, remifentanil was administered last after the propofol and rocuronium injection
  Interventions: Drug: the order of drug administration

INTERVENTIONS:
Drug: the order of drug administration — In group R, remifentanil was infused first before administrating propofol and rocuronium and in group P, it was administered last after the rocuronium injection. In other words, the order of drug infusion in each group is remifentanil-propofol-rocuronium in group R and propofol-rocuronium-remifentanil in group P, respectively.
  Other Names: esmeron; ultiva; fresopol

SUMMARY:
The investigators therefore hypothesized that remifentanil could prolong the onset time of rocuronium, and evaluated the effect of remifentanil on the hemodynamic profiles (arterial pressure and heart rate) during the anesthetic induction sequence.

DETAILED DESCRIPTION:
It has been reported that co-administration of ephedrine reduced the onset time of neuromuscular block of rocuronium (1-3). It also provided an improved condition for the rapid tracheal intubation (2,4). This beneficial effect was attributed to the increased cardiac output and tissue perfusion to muscle, and therefore, a more rapid delivery of rocuronium to the neuromuscular junction was achieved (4-5). If so, any drugs which decrease cardiac output consequently can prolong the onset time of rocuronium.

Remifentanil is the first ultra-short acting opioid with a rapid onset. During the total intravenous anesthesia (TIVA) with propofol and remifentanil, prior administration of remifentanil could reduce the propofol infusion pain without other significant complications (6). However, remifentanil can decrease the arterial pressure and heart rate (7-8), so that it is likely to decrease the onset time of rocuronium for the opposite principle that ephedrine increases it.

The investigators therefore hypothesized that remifentanil could prolong the onset time of rocuronium, and evaluated the effect of remifentanil on the hemodynamic profiles (arterial pressure and heart rate) during the anesthetic induction sequence.

ELIGIBILITY:
Inclusion criteria:

* American Society of Anesthesiologist physical status I or II
* Aged 20-65 yr
* Elective surgery under general anesthesia with total intravenous anesthesia
* 8.5 kg/m2 < body mass index (BMI) < 25 kg/m2

Exclusion criteria:

* BMI > 25 kg/m2 or < 18.5 kg/m2
* Any cardiovascular or neuromuscular disease
* Intake of drugs known to interact with the neuromuscular junction
* Patients wit risk of pulmonary aspiration
* Anticipated difficult airway
* history of known allergy to rocuronium

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
the onset time of rocuronium | 3 minutes [after injection of rocuronium when general anesthesia is induced.]
  Onset time of rocuronium was defined as the time from the end of its injection to the 95% depression of single twitch response, and it was measured by an anaesthesiologist, unaware of the group allocation.

SECONDARY OUTCOMES:
mean arterial pressure (MAP) | 15 minutes [4 times; during the induction of general anesthesia as described below.]
  1. before induction (baseline): When a patient enter the operating room,
  2. at rocuronium administration: immediately before injecting rocuronium,
  3. before tracheal intubation: immediately before intubation,
  4. after tracheal intubation: immediately after intubation.
heart rate (HR) | 15 minutes [4 times; during the induction of general anesthesia as described below.]
  1. before induction (baseline): When a patient enter the operating room,
  2. at rocuronium administration: immediately before injecting rocuronium,
  3. before tracheal intubation: immediately before intubation,
  4. after tracheal intubation: immediately after intubation.
cardiac output | 15 minutes [4 times; during the induction of general anesthesia as described below.]
  1. before induction (baseline): When a patient enter the operating room,
  2. at rocuronium administration: immediately before injecting rocuronium,
  3. before tracheal intubation: immediately before intubation,
  4. after tracheal intubation: immediately after intubation.
pain from the propofol infusion | 1 minute [at the time when propofol is administered.]
  When propofol is administered for the induction of anesthesia, we investigate the pain by propofol.
cough or chest wall rigidity from the remifentanil infusion | 1 minute [at the time when remifentanil is infused.]
  when remifentanil is infused, the cough or chest wall rigidity is checked.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea